CLINICAL TRIAL: NCT01682928
Title: Submersion Therapy for the Reversal of Oligohydramnios; A Non-invasive Gentle Approach
Brief Title: Hydrotherapy for the Reversal of Oligohydramnios
Acronym: STRONG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Pediatrix (Other)
Collaborators: Banner Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRONG-2012
Record Dates: First submitted 2012-09-06; First posted 2012-09-11 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Oligohydramnios
Keywords: Oligohydramnios; Hydrotherapy; Pregnancy
MeSH Terms: conditions — Oligohydramnios | interventions — Bed Rest; Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV/Oral Hydration and Bedrest (Active Comparator): * Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
  Interventions: Drug: IV/Oral Hydration and Bedrest
- Hydrotherapy Group (Active Comparator): * Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
    o 1 hour +/- 30 minutes after submersion therapy
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
    o 1 hour +/- 30 minutes after submersion therapy
  * AFI (Baseline, day 3, 7 {or Discharge}) o 1 hour +/- 30 minutes after submersion therapy
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
  * HYDROTHERAPY TWICE DAILY FOR 3-7 DAYS o Blood pressure, pulse, pulse pressure, body weight, and fetal heart rate before and after submersion therapy
  Interventions: Other: Hydrotherapy

INTERVENTIONS:
Drug: IV/Oral Hydration and Bedrest — * Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
  Arms: IV/Oral Hydration and Bedrest
Other: Hydrotherapy — * Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
    o 1 hour +/- 30 minutes after submersion therapy
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
    o 1 hour +/- 30 minutes after submersion therapy
  * AFI (Baseline, day 3, 7 {or Discharge}) o 1 hour +/- 30 minutes after submersion therapy
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
  * HYDROTHERAPY TWICE DAILY FOR 3-7 DAYS o Blood pressure, pulse, pulse pressure, body weight, and fetal heart rate before and after submersion therapy
  Arms: Hydrotherapy Group

SUMMARY:
OBJECTIVE: To assess the efficacy of subtotal immersion therapy as an option to improve maternal intravascular volume thereby improving both maternal and fetal hemodynamic status with reversal of oligohydramnios. This will be measured utilizing the Amniotic Fluid Volume (AFV) as the primary outcome. Secondary outcomes will be measured using Fetal Doppler Studies, Maternal vital signs (Blood Pressure, Pulse Pressure, Weight, Pulse) and input/output.

HYPOTHESIS: Oligohydramnios, secondary to depleted maternal intravascular volume, can be reversed by improving feto- and uteroplacental perfusion with subtotal immersion therapy.

DETAILED DESCRIPTION:
BACKGROUND: The volume of amniotic fluid is relevant clinically as derangements that decrease volume result in a condition known as oligohydramnios, which can have profound implications on perinatal outcome. The incidence of oligohydramnios is 2.3%1,2,3 and measurements of amniotic fluid volume (AFV) has become a standard in fetal surveillance in the evaluation of high risk pregnancies as oligohydramnios is associated with intrauterine growth restriction, respiratory distress syndrome, post-maturity syndrome, and chronic fetal hypoxia. Oligohydramnios may also play a role in fetal malpresentation, umbilical cord compression, meconium staining, and increased operative delivery.3,4, 5,6 Oligohydramnios is commonly defined as an AFV of 5 cm or less. An AFV of 8 cm represents the fifth percentile of normal AFV values.7 It has been observed that delivery in the setting of isolated oligohydramnios, irrespective of an otherwise uncomplicated term gestation free of maternal disease, has become routine thereby increasing maternal morbidity particularly in context of operative delivery or failed inductions. 3

In order to understand oligohydramnios it is first important to understand intrauterine water and progressive changes that occur with normal human gestation. At term, it is reported that total water accumulation is approximately 3.5L, with 2400 mL in the fetus, 400 mL in the placenta, and 700 mL in the amniotic fluid.8 In 1989, Brace and colleagues determined amniotic fluid volume (AFV) as a function of gestational age. They reported an increase in mean values from 30mL at 10weeks to 190mL at 16wks to 780mL at 32-35wks after which time AFV decreases, especially in post-term pregnancies. It is important to realize; however, that the pattern of volume fluctuation as a function of gestational age may vary considerably between individuals. As a general rule AFV increases at a rate of 10ml/wk at the beginning of the fetal period, this rate of expansion increases to 50-60ml/wk from 19 to 25wks at which time a gradual decrease begins to take place until the rate of exchange is zero around 34wks.

The pathophysiology of amniotic fluid regulation is not entirely understood at this current date, but it is safe to state that AFV is the integrated sums of the inflow and outflow tracts of the amniotic space.8 Because fluid can move with relative ease between fetal and maternal blood across the placenta and amniotic membranes it stands to reason that a maternal hypovolemia secondary to dehydration would lead to the development of oligohydramnios. This was indeed shown to be the case by Sherer, et al in their 1990 publication. Furthermore, both oral and serum hydration as a way to increase maternal volume have been shown to be effective treatments for oligohydramnios.3,11-16

ELIGIBILITY:
Inclusion Criteria:

* Maternal Age >18 years
* Oligohydramnios: diagnosed by sonography (defined AFV<8cm)
* Singleton Pregnancy
* Intact membranes
* Gestational age 24 - 36 weeks

Exclusion Criteria:

* Indication for urgent delivery (severe PET, HELLP syndrome, persistent fetal hypoxemia [non-reassuring fetal heart rate pattern])
* Ruptured amniotic membranes; PPROM, PROM, SROM
* Fever (>38C)
* Multiple gestation
* >37 week gestation
* Lethal Fetal anomalies and/or demise
* Maternal Cardiovascular disease
* Maternal Renal disease
* Maternal Pulmonary disease (other than asthma)
* Patients using prostaglandin inhibitors, NSAIDs3,15 (within 1 week of enrollment, other than baby asprin)
* Non-English speaking
* Vaginal Infections and/or active skin lesions
* Placenta Previa and/or Unexplained Vaginal Bleeding
* BMI > 45

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Strong, MD, Principal Investigator — Obstetrix Medical Group
Locations (1):
- Banner Good Samaritan Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began April 8, 2012 and ended April 2014. Recruitment took place at Banner Good Samaritan hospital based on Banner IRB approval.
Pre-assignment Details: There were no pre-assignment events.
Groups:
- IV/Oral Hydration and Bedrest: 1 Liter Water PO over 2 hours
  1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation Strict I/O's Vital signs US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
- Hydrotherapy Group: US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline,
  * Uterine Artery Doppler Flow (Baseline,
  * AFI (Baseline,
  * Strict I/O's
  * Vital signs
  * HYDROTHERAPY TWICE DAILY FOR 3-7 DAYS
    o Blood pressure, pulse, pulse pressure, body weight, and fetal heart rate before and after submersion therapy Hydrotherapy: • Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow
  * Uterine Artery Doppler Flow • AFI (Baseline, day 3, 7 {or Discharge})
Period: Overall Study
Arm/Group | IV/Oral Hydration and Bedrest | Hydrotherapy Group
Started | 2 (2 subjects in this Arm) | 2 (2 subjects in this Arm)
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hydrotherapy Group: • HYDROTHERAPY TWICE DAILY FOR 3-7 DAYS
  o Blood pressure, pulse, pulse pressure, body weight, and fetal heart rate before and after submersion therapy
  Hydrotherapy:
  * Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
    o 1 hour +/- 30 minutes after submersion therapy
  * AFI (Baseline, day 3, 7 {or Discharge}) o 1 hour +/- 30 minutes after submersion therapy
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
- Total: Total of all reporting groups
Arm/Group | IV/Oral Hydration and Bedrest | Hydrotherapy Group | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 31.5 [29 to 34] | 23 [21 to 25] | 27.25 [21 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 1. Primary: Number of Participants With Reversal of Oligohydramnios Using AFV Measures
Description: Subjects amniotic fluid index via ultrasound on days 3, 5 and 7 of study participation.
Time Frame: days 3, and 7 or discharge
Population: no formal analysis done on the 4 enrolled patients, study halted due to poor enrollment. Data cannot be reported due to participant privacy.
Groups:
- IV/Oral Hydration and Bedrest: IV/Oral Hydration and Bedrest for up to 7 days
  US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
    : • Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV
- Hydrotherapy Group: HYDROTHERAPY TWICE DAILY FOR 3-7 DAYS
  * Maternal BP (sitting) US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
    o 1 hour +/- 30 minutes after submersion therapy
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
    o 1 hour +/- 30 minutes after submersion therapy
  * AFI (Baseline, day 3, 7 {or Discharge}) o 1 hour +/- 30 minutes after submersion therapy
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
    * Blood pressure, pulse, pulse pressure, body weight, and fetal heart rate before and after submersion therapy
  Hydrotherapy: • Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight
Arm/Group | IV/Oral Hydration and Bedrest | Hydrotherapy Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Metabolic Status
Description: Secondary:
  - Changes in maternal hemodynamic status by mobilizing extravascular fluid
Time Frame: admission, days 3, 5, 7/discharge and delivery
Population: No analysis done as study halted for poor enrollment only 4 subjects enrolled total. Detailed Data cannot be reported due to participant privacy.
Groups:
- IV/Oral Hydration and Bedrest: IV/Oral Hydration and Bedrest up to 7 days
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
    : • Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital sign
- Hydrotherapy Group: • HYDROTHERAPY TWICE DAILY FOR 3-7 DAYS
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
    * Blood pressure, pulse, pulse pressure, body weight, and fetal heart rate before and after submersion therapy
  Hydrotherapy: • Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge}) o 1 hour +/- 30 minutes after submer
Arm/Group | IV/Oral Hydration and Bedrest | Hydrotherapy Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years and 4 months
Groups:
- IV/Oral Hydration and Bedrest: * Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
  ALL ITEMS ABOVE MUST BE COMPLETED BEFORE:
  * 1 Liter Water PO over 2 hours
  * 1 Liter IV Fluid Bolus (NS) then titrated to 75 ml\hr for duration of the study participation
  * Strict I/O's
  * Vital signs
  IV/Oral Hydration and Bedrest: • Maternal BP (sitting)
  * Pulse Pressure
  * Pulse
  * Urine Specific Gravity BID
  * Fetal Heart Rate
  * Maternal Body Weight US Procedures
  * AC/EFW
  * Umbilical Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * Uterine Artery Doppler Flow (Baseline, day 3, 7 {or Discharge})
  * AFI (Baseline, day 3, 7 {or Discharge})
Arm/Group | IV/Oral Hydration and Bedrest | Hydrotherapy Group
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No